CLINICAL TRIAL: NCT06799845
Title: A Phase 2B, Randomized, Double Blind, Placebo and Active Comparator Controlled, Multicenter, Safety, and Efficacy Trial of ATX101 in Adults Undergoing Total Knee Arthroplasty
Brief Title: Study Assessing Pain Relief After Replacement of the Knee
Acronym: SPARK 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX-101-TKA-004
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Total Knee Arthroplasty (Postoperative Pain)
Keywords: postoperative pain; post-surgical pain total knee arthroplasty; bupivacaine; bupivacaine implant; total knee replacement; ATX101; TKA; post-operative pain; postsurgical pain; post-surgical pain; postsurgical pain total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: surgical staff and pharmacist dispensing assigned treatment will not be blinded to the trial treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATX101 (Experimental)
  Interventions: Drug: ATX101
- saline placebo (Placebo Comparator)
  Interventions: Drug: saline placebo
- bupivacaine hydrochloride (Active Comparator)
  Interventions: Drug: bupivacaine hydrochloride

INTERVENTIONS:
Drug: ATX101 — ATX101 bupivacaine implants, total of 1,500 mg into the surgical site
  Arms: ATX101
Drug: bupivacaine hydrochloride — bupivacaine hydrochloride 0.25% without epinephrine/adrenaline, total 125 mg in 50 mL via local periarticular infiltration
  Arms: bupivacaine hydrochloride
Drug: saline placebo — normal saline (0.9%) sodium chloride, total volume of up to 17 mL via local periarticular infiltration
  Arms: saline placebo

SUMMARY:
The goal of the ATX101-TKA-004 clinical trial aims to evaluate the efficacy and safety of ATX101 1,500 mg in participants undergoing primary unilateral total knee arthroplasty. The study will compare the effectiveness of ATX101 with a saline placebo and bupivacaine, an active comparator. Additionally, it will assess opioid consumption among participants receiving ATX101 versus those given the saline placebo and bupivacaine. The trial will also focus on the safety and tolerability of ATX101 in the participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Primary indication of TKA is knee pain due to osteoarthritis or post-traumatic arthritis
* Scheduled to undergo primary unilateral TKA with a cemented prosthesis, without use of a surgical drain, and under bupivacaine spinal anesthesia (dextrose is permitted)
* American Society of Anesthesiology (ASA) Physical Classification System of class 1, 2, or 3
* Capable, able, and willing to comply with all trial visits and procedures. Participant must also be able to use trial required e-diary and demonstrate completion compliance during the screening period
* English or Spanish speaking, willing, and capable of providing written informed consent

Key Exclusion Criteria:

* Has a planned concurrent surgical procedure (e.g. bilateral TKA) at the time of surgery or a planned surgical procedure before the last trial visit
* Has had any previous open surgery, (e.g., ORIF for fracture, osteotomy, arthroplasty, unicompartmental knee arthroplasty, or TKA), in the trial knee at any time in the past or arthroscopic surgery within 12 months. Has had any previous surgery in the contralateral knee within 6 months prior to screening
* Has been administered any type of intra-articular injection within 3 months of surgery in the trial knee
* Unable to abstain from opioid use for knee pain (including codeine) within 2 weeks (14 days) of surgery
* Has a Body Mass Index (BMI) ≥45 kg/m²
* Is unwilling or unable to discontinue use of medications or products that can impact pain control from the Screening Visit until the last trial visit (e.g. cannabidiol (CBD) oil, Kratom)
* Has a medical condition or receiving medication such that, in the opinion of the Investigator, participating in the trial would pose a health risk to the participant or confound the postsurgical assessments or might confound or interfere with the outcome of the trial
* Has received/used an investigational drug, product, or device for a clinical trial within 30 days of screening. COVID-19 vaccines (approved or under emergency use authorization locally) are permitted if the participant is not in a clinical trial for the vaccine
* Has a positive drug screen at the Screening Visit or on the day of surgery
* Has participated in an ATX101 clinical trial
* Pregnant, breastfeeding, or planning to become pregnant during the trial or before the last trial visit

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for the Numerical Rating Scale at Rest (NRS-R) of pain intensity | from 30 minutes through 168 hours (Day 8) compared to placebo
  NRS-R for pain intensity is an 11-item scale from 0 to10 where participants rank the level of pain intensity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).

SECONDARY OUTCOMES:
AUC for the NRS-R of pain intensity | 30 minutes through 336 hours (Day 15) compared to placebo
  NRS-R for pain intensity is an 11-item scale from 0 to10 where participants rank the level of pain intensity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).
AUC for the NRS-R of pain intensity | from 30 minutes through 504 hours (Day 22) compared to placebo
  NRS-R for pain intensity is an 11-item scale from 0 to10 where participants rank the level of pain intensity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).
Total post-surgical consumption of opioid medications | from 30 minutes through 336 hours (Day 15) compared to placebo
AUC for the NRS-R of pain intensity | from 30 minutes through 336 hours (Day 15) compared to active comparator
  NRS-R for pain intensity is an 11-item scale from 0 to10 where participants rank the level of pain intensity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).
Difference in NRS-A pain intensity scores during the Timed Up and Go (TUG) Test | at Day 15 compared to placebo
  The NRS with activity (NRS-A) for pain intensity is an 11-item scale from 0 to 10 where participants rank the level of pain intensity after an activity. The NRS scale goes from No Pain (0) to Worst Imaginable Pain (10).

CONTACTS AND LOCATIONS:
Overall Officials: David Hewitt, MD, Study Director — Allay Therapeutics, Inc.
Locations (11):
- United States (11):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Phoenix Clinical Research, Tamarac, Florida
  - Atlanta Centre for Medical Research, Atlanta, Georgia
  - NextStage Clinical Research, Wichita, Kansas
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - Memorial Hermann Village, Houston, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - NextStage Clinical Research, San Antonio, Texas
  - JBR Clinical Research, LLC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No